CLINICAL TRIAL: NCT05308628
Title: Effect of the Fibrosis Panel on the Evaluation of Allograft Fibrosis After Pediatric Liver Transplantation
Brief Title: Pediatric Liver Transplantation-Liver Fibrosis Evaluation by Using Fibrosis Panel
Acronym: PT-LiFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Renji-IIT-2022-0002
Record Dates: First submitted 2022-01-17; First posted 2022-04-04 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Liver Fibrosis; Pediatric Disorder; Liver Transplant; Complications
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-Transplant-Liver Allograft Fibrosis (Active Comparator): Pediatric patients who have undergone liver transplantation , the occurrence of graft fibrosis necessitates hospitalization for biopsy and treatment to assess the degree of fibrosis and its underlying causes.
  Interventions: Diagnostic Test: Liver Allograft Fibrosis by Using Fibrosis Panel(PRO-C3, PIIINP, TIMP-1, HA etc.)
- Post-Transplant-Liver Allograft regular recovery (Sham Comparator): Pediatric patients who have undergone liver transplantation and have recovered normally typically undergo liver biopsy around 3 to 5 years postoperatively and around 10 years postoperatively to evaluate the presence of potential subclinical rejection. This assessment guides the long-term application of immunosuppressive medications.
  Interventions: Diagnostic Test: Liver Allograft Fibrosis by Using Fibrosis Panel(PRO-C3, PIIINP, TIMP-1, HA etc.)

INTERVENTIONS:
Diagnostic Test: Liver Allograft Fibrosis by Using Fibrosis Panel(PRO-C3, PIIINP, TIMP-1, HA etc.) — Liver biopsies will be performed at 3 months, 6 months and 12 months post-transplant. Fibrosis was evaluated using the liver allograft fibrosis score (LAFSc) staging system. Liver Allograft Fibrosis by Using Fibrosis Panel(PRO-C3, PIIINP, TIMP-1, HA)or (FBLN3,YKL40,LECT2 etc.)
  Other Names: Liver Allograft Fibrosis by Using Fibrosis Panel(FBLN3,YKL40,LECT2 etc.)

SUMMARY:
Liver transplantation in children is highly successful with >80% having 20 years survival. Most pediatric liver diseases are potentially curable with liver transplantation and it is important to establish whether children who have undergone successful transplantation can expect a normal life expectancy or whether there will be a gradual decline in liver function and eventual graft loss. The most common reasons in late graft loss in children are unexplained graft inflammation ("idiopathic" post-transplant hepatitis) and graft fibrosis. PRO-C3, a disintegrin and metalloproteinase with thrombospondin motifs-generated neo-epitope marker of type III collagen formation, has been proved to be a marker of fibrosis in patients with NAFLD. The aim of this study is to explore the role of Fibrosis Panel(PRO-C3, PIIINP, TIMP-1, HA) in children received liver transplantation.

DETAILED DESCRIPTION:
The cross-section study will be performed in pediatric patients who underwent liver transplantation from year 2016-2021. Patients will be enrolled after collecting their informed consent from their parents. As soon as the patient is included, arrangements will be made for the liver biopsy according to the schedule.

Liver biopsies will be performed at 3 months, 6 months and 12 months post-transplant. For the purpose of this study, each section was independently and blindly reassessed by expert pathologists. Fibrosis was evaluated using the liver allograft fibrosis score (LAFSc) staging system [Fibrosis deposition was classified in three main areas of the liver parenchyma: portal tracts, sinusoids (zones 1 and 2) and centrolobular veins (zone 3); in each area, fibrosis was staged from 0 to 3 (0 = absent, 1 = mild, 2 = moderate and 3 = severe fibrosis), with a total score of 9. Equal score weight was assigned to each area] and the Ishak staging system (0 = no fibrosis; 1 = fibrous expansion of some portal area; 2 = fibrous expansion of most portal areas; 3 = fibrous expansion of most portal areas with occasional bridging; 4 = fibrous expansion of most portal areas with marked bridging; 5 = marked bridging occasional nodules; and 6 = cirrhosis).

At the time of biopsy, a fasting blood sample was obtained and routine biochemical tests were performed using standard methods and assays. Additional blood samples were drawn and frozen at -80℃ for future research. Type III collagen formation was assessed in serum using the Fibrosis Panel(PRO-C3, PIIINP, TIMP-1, HA) competitive enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant must be between 8 weeks and 18 years of age.
* Participant is a recipient of a first liver allograft from cadaveric or living donors.
* Participant is a single-organ recipient (liver only).
* Participants' parent/guardian is capable of understanding the purposes and risks of the study and must sign an informed consent for the study.

Exclusion Criteria:

* Participants older than 18 years of age
* Pregnant or breastfeeding
* Active systemic infections
* Receiving any form of solid organ retransplantation
* Multiorgan transplantation
* Multi organ failure
* Congenital sufferers from heart, lung, kidney, nervous system or blood disease
* Refused to participate the study

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
liver allograft fibrosis score (LAFSc) staging system(12 months) | 12 months post-transplant
  Fibrosis deposition was classified in three main areas of the liver parenchyma: portal tracts, sinusoids (zones 1 and 2) and centrolobular veins (zone 3); in each area, fibrosis was staged from 0 to 3 (0 = absent, 1 = mild, 2 = moderate and 3 = severe fibrosis), with a total score of 9. Equal score weight was assigned to each area] and the Ishak staging system (0 = no fibrosis; 1 = fibrous expansion of some portal area; 2 = fibrous expansion of most portal areas; 3 = fibrous expansion of most portal areas with occasional bridging; 4 = fibrous expansion of most portal areas with marked bridging; 5 = marked bridging occasional nodules; and 6 = cirrhosis

SECONDARY OUTCOMES:
liver allograft fibrosis score (LAFSc) staging system(6 months) | 6 months post-transplant
  Fibrosis deposition was classified in three main areas of the liver parenchyma: portal tracts, sinusoids (zones 1 and 2) and centrolobular veins (zone 3); in each area, fibrosis was staged from 0 to 3 (0 = absent, 1 = mild, 2 = moderate and 3 = severe fibrosis), with a total score of 9. Equal score weight was assigned to each area] and the Ishak staging system (0 = no fibrosis; 1 = fibrous expansion of some portal area; 2 = fibrous expansion of most portal areas; 3 = fibrous expansion of most portal areas with occasional bridging; 4 = fibrous expansion of most portal areas with marked bridging; 5 = marked bridging occasional nodules; and 6 = cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Hao FENG, Study Director — Dept. of Liver surgery, Renji Hospital, Medical School of Shanghai Jiaotong University
Locations (2):
- China (2):
  - Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai
  - Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai